CLINICAL TRIAL: NCT03670251
Title: Improving Access to Viral Load Monitoring in HIV-infected Patients on ART in Decentralised Area Using Dried Blood Spot : Evaluation of Hepatitis C Viral Load Quantification on DBS
Brief Title: Evaluation of Hepatitis C Viral Load Quantification on DBS in Vietnam
Acronym: MOVIDA-Hep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Hanoi University of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-076
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C; Dried Blood Spot
Keywords: HCV Viral Load, Dried Blood Spot, HCV Core Ag
MeSH Terms: conditions — Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Other): blood samples from venepuncture (10mL) and from fingertip (approximatively 0.4mL) on a dried blood spots
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sample of 10 mL by venipuncture and 0,4 mL by finger prick

SUMMARY:
In Vietnam, the prevalence of hepatitis C virus (HCV) infection is estimated between 0.4% and 5%, which is much higher than the prevalence in Europe or in the USA. After HCV diagnosis, HCV viral load quantification is crucial in order to distinguish recovered from active (on-going) HCV infection and hence identify those who need antiviral treatment to cure HCV infection. HCV viral load quantification is also important to assess treatment efficacy.

Currently, anti-HCV antibodies detection is available around the country. However, access to confirmation of HCV viremia remains scarce particularly in decentralized areas. One of the reason is the limited number of laboratories able to perform this complex biological measurement; moreover, these laboratories are situated only in large urban centres.

Blood sampling using DBS could help overcome this difficulty of access to a laboratory, and widen access to HCV viral load monitoring.

The present MOVIDA Hep study aims at validating the use of DBS to measure HCV viral load as compared to plasma (gold standard). A secondary objective is to evaluate the measurement of HCV core antigen on DBS. For this, 315 patients need to be enrolled form outpatient clinics in Hanoi. The laboratory in charge of these measurements would be the virology laboratory of the National Institute of Hygiene and Epidemiology (NIHE) in Hanoi (Vietnam).

DETAILED DESCRIPTION:
The "Monitoring Of Viral load In Decentralised Area" (MOVIDA) project aims at giving access to viral load (VL) monitoring to the patients coming from remote areas using Dried Blood Spot as tool of sampling.

In resource-limited settings, many biological exams are not accessible to the entire population due to logistic and financial constraints. Regarding infection with hepatitis B and C viruses (HBV and HCV), serological screening tests are easy to perform and are available nationwide in either laboratory format or rapid diagnosis tests. However, hepatitis B DNA and C RNA assessment is not available in decentralised area as no laboratory is able to perform this complex biological measurement.

WHO, in their latest guidelines, recommends using dried blood spots (DBS) as an alternative to serum or plasma. Blood is easy to collect on DBS, either after veni- or capillary puncture. Capillary blood collection can be of great interest when venipuncture is complex, for example in injecting drug users (IDUs) in whom finding an accessible vein can be difficult. Then it is easily transferred, and at a low cost as it does not require a cold chain, to a laboratory able to perform the HCV VL quantification. As of today, little is known about the performance of standard commercial HCV diagnostic assays when using DBS and none of these studies were performed in routine setting in resource-limited setting.

In Vietnam, HCV seroprevalence in the general population is estimated between 0.4% and 5%, which is much higher than the prevalence in Europe or in the US. Genotype 1 is the more prevalent in Vietnam, genotype 6 that is only found in South East Asia is the second most frequent, but other genotypes are circulating . In Vietnam, HCV prevalence is much higher in the HIV-infected population and in injecting drug users (IDUs). Currently, anti-HCV antibodies detection is available around the country even if some difficulties remain. However, access to HCV HCV viral load measurement in routine remains scarce particularly in decentralized areas because the technique is complex, expensive and need well-trained personnel and high standard of equipment. Thus, HCV viral load measurement remains non accessible to the vast majority of patients diagnosed with HCV.

This study (MOVIDA Hep) aims at evaluating the quality of HCV VL monitoring when using DBS (collection of venous and capillary blood) as compared to plasma (gold standard), in routine condition and using the existing machines. This, to find out if DBS can be used for HCV viremia confirmation in Vietnam, in the virology laboratory of the National Institute of Hygiene and Epidemiology (NIHE) in Hanoi (Vietnam) where these measurements would be performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Known HCV infection
* Willing to participate to the study by giving his/her consent.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Quantification of HCV RNA on DBS compared to plasma as gold standard | Up to 4 weeks
  Sensitivity and specificity of HCV RNA VL measured on DBS collected by venipuncture

SECONDARY OUTCOMES:
Quantification of HCV RNA measured on DBS using plasma as gold standard | Up to 4 weeks
  Sensitivity and specificity of HCV RNA VL measured on DBS collected by finger prick
Correlation between HCV RNA VL measured on DBS and on plasma. | Up to 6 months
  Correlation between HCV RNA VL measured on DBS (collected by venipuncture and finger prick) and on plasma.
Quantification of HCV core antigen using HCV RNA VL as gold standard | Up to 8 weeks
  Sensitivity and specificity of HCV core antigen using HCV RNA VL as gold standard
Correlation between HCV core antigen and HCV RNA VL on plasma | Up to 6 months
  Correlation between HCV core antigen and HCV RNA VL, both measured on plasma.
Quantification of HCV core antigen measured on DBS using HCV RNA VL measured on plasma as gold standard. | Up to 8 weeks
  Sensitivity and specificity of HCV core antigen measured on DBS collected by venipuncture using HCV RNA VL measured on plasma as gold standard.
Correlation between HCV core antigen measured on DBS and HCV RNA VL measured on plasma. | Up to 6 months
  Correlation between HCV core antigen measured on DBS collected by venipuncture and HCV RNA VL measured on plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien TAIEB, MD, PhD, MPH, Principal Investigator — Institut Pasteur; Tuan Anh NGUYEN, MD, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology (NIHE)
Locations (2):
- Vietnam (2):
  - Dong Da Hospital, Hanoi
  - Nam Tu Liem Hospital, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taieb F, Tran Hong T, Ho HT, Nguyen Thanh B, Pham Phuong T, Viet Ta D, Le Thi Hong N, Ba Pham H, Nguyen LTH, Nguyen HT, Nguyen TT, Tuaillon E, Delaporte E, Le Thi H, Tran Thi Bich H, Nguyen TA, Madec Y. First field evaluation of the optimized CE marked Abbott protocol for HIV RNA testing on dried blood spot in a routine clinical setting in Vietnam. PLoS One. 2018 Feb 9;13(2):e0191920. doi: 10.1371/journal.pone.0191920. eCollection 2018. PMID 29425216
- [Background] Taieb F, Tram TH, Ho HT, Pham VA, Nguyen L, Pham BH, Tong LA, Tuaillon E, Delaporte E, Nguyen AT, Bui DD, Do N, Madec Y. Evaluation of Two Techniques for Viral Load Monitoring Using Dried Blood Spot in Routine Practice in Vietnam (French National Agency for AIDS and Hepatitis Research 12338). Open Forum Infect Dis. 2016 Jul 7;3(3):ofw142. doi: 10.1093/ofid/ofw142. eCollection 2016 Sep. PMID 27704001
- [Background] Soulier A, Poiteau L, Rosa I, Hezode C, Roudot-Thoraval F, Pawlotsky JM, Chevaliez S. Dried Blood Spots: A Tool to Ensure Broad Access to Hepatitis C Screening, Diagnosis, and Treatment Monitoring. J Infect Dis. 2016 Apr 1;213(7):1087-95. doi: 10.1093/infdis/jiv423. Epub 2015 Sep 2. PMID 26333945
- [Result] Tran TH, Nguyen BT, Nguyen TA, Pham TTP, Nguyen TTT, Mai HTB, Pham HB, Nguyen TM, Phan HTT, Do NT, Ait-Ahmed M, Taieb F, Madec Y. Dried blood spots perform well to identify patients with active HCV infection in Vietnam. J Viral Hepat. 2020 May;27(5):514-519. doi: 10.1111/jvh.13263. Epub 2020 Feb 11. PMID 31981287
- See also: WHO Guidelines on Hepatitis B and C Testing — http://apps.who.int/iris/bitstream/10665/254621/1/9789241549981-eng.pdf